CLINICAL TRIAL: NCT00791661
Title: A Single Dose Clinical Trial to Study the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of MK-1006 in Japanese Subject With Type 2 Diabetes
Brief Title: MK-1006 Single Dose Study in Japanese Type 2 Diabetes Patients (MK-1006-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1006-005; 2008_584
Record Dates: First submitted 2008-11-10; First posted 2008-11-14 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A: MK-1006 15/30/45 (Experimental): Participants received a single rising dose of MK-1006 (dosed at 15 mg, 30 mg, and 45 mg) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
  Interventions: Drug: MK-1006; Drug: Placebo
- Panel B: MK-1006 60/80/60 fed (Experimental): Participants received a single rising dose of MK-1006 (dosed at 60 mg, 80 mg, and 60 mg fed state) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
  Interventions: Drug: MK-1006; Drug: Placebo
- Panel C: MK-1006 100/140/170 (Experimental): Participants received a single rising dose of MK-1006 (dosed at 100 mg, 140 mg, and 170 mg) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
  Interventions: Drug: MK-1006; Drug: Placebo

INTERVENTIONS:
Drug: MK-1006 — MK-1006 capsules in single oral doses beginning at 15 mg and rising to 45 mg in Panel A, beginning at 60 mg and rising to 80 mg and 60 mg fed state in Panel B, or beginning at 100 mg and rising to 170 mg in Panel C.
Drug: Placebo — Matching placebo to MK-1006 in a single oral dose

SUMMARY:
A single rising dose study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of MK-1006 in Japanese participants with Type 2 Diabetes Mellitus (T2DM). The primary hypothesis of the study is that single doses of MK-1006 will be sufficiently safe and well tolerated, based on the assessment of clinical and laboratory evaluations and adverse experiences, in Japanese participants with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female between 20 to 64 years of age
* Diagnosis of type 2 diabetes
* Patient is being treated with diet and exercise alone or single oral anti-hyperglycemic agent

Exclusion Criteria:

* Subject has a history of type 1 diabetes mellitus
* Subject has a clinical diagnosis of glaucoma
* Subject has donated blood or participated in another clinical study in the past 12 weeks
* Subject is a regular user of any illicit drugs or has a history of drug, including alcohol, abuse in the past 6 months

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A: MK-1006 15/30/45: Participants received a single dose of MK-1006 (dosed at 15 mg, 30 mg, and 45 mg) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
- Panel B: MK-1006 60/80/60 Fed: Participants received a single dose of MK-1006 (dosed at 60 mg, 80 mg, and 60 mg fed state) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
- Panel C: MK-1006 100/140/170: Participants received a single dose of MK-1006 (dosed at 100 mg, 140 mg, and 170 mg) or matching placebo to MK-1006 with a 7-day wash-out period between doses. Participants could have received both MK-1006 and matching placebo to MK-1006 over the 3 treatment periods.
Period: Period 1
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170
Started | 8 | 8 | 8
Received MK-1006 | 6 | 6 | 6
Received Matching Placebo to MK-1006 | 2 | 2 | 2
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: 7 Day Wash-out
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170
Started | 8 | 8 | 8
Completed | 8 | 8 | 6
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Abnormal Clinical Laboratory Test | 0 | 0 | 1
Period: Period 2
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170
Started | 8 | 8 | 6
Received MK-1006 | 6 | 6 | 4
Received Matching Placebo to MK-1006 | 2 | 2 | 2
Completed | 8 | 8 | 6
Not Completed | 0 | 0 | 0
Period: 7 Day Wash-out
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170
Started | 8 | 8 | 6
Completed | 8 | 8 | 6
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170
Started | 8 | 8 | 6
Received MK-1006 | 6 | 6 | 5
Received Matching Placebo to MK-1006 | 2 | 2 | 1
Completed | 8 | 8 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-1006 15/30/45 | Panel B: MK-1006 60/80/60 Fed | Panel C: MK-1006 100/140/170 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Customized [Number; unit: Participants]
  <41 years | 0 | 0 | 0 | 0
  >= 41 years and <=64 years | 8 | 8 | 8 | 24
  >64 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 8 | 5 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Japan | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Time Frame: from the time of the run-in period prior to the first dose of study drug through the end of the poststudy period (up to approximately 31 days)
Population: Participants who received study drug. The same participant may appear in more than one treatment arm.
Measure: Number; unit: participants
Groups:
- MK-1006 15 mg: Participants received a single dose of MK-1006 15 mg
- MK-1006 30 mg: Participants received a single dose of MK-1006 30 mg
- MK-1006 45 mg: Participants received a single dose of MK-1006 45 mg
- MK-1006 60 mg: Participants received a single dose of MK-1006 60 mg
- MK-1006 60 mg Fed: Participants received a single dose of MK-1006 60 mg following consumption of a standard Japanese breakfast
- MK-1006 80 mg: Participants received a single dose of MK-1006 80 mg
- MK-1006 100 mg: Participants received a single dose of MK-1006 100 mg
- MK-1006 140 mg: Participants received a single dose of MK-1006 140 mg
- MK-1006 170 mg: Participants received a single dose of MK-1006 170 mg
- Placebo: Participants received matching placebo to MK-1006
- Placebo Fed: Participants received matching placebo to MK-1006 following consumption of a standard Japanese breakfast
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg | Placebo | Placebo Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5 | 15 | 2
participants | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 1 | 1

2. Secondary Outcome: Mean Area Under the Plasma Concentration Curve From Time Zero to Infinity(AUC[0-∞]) After a Single Dose of MK-1006
Description: AUC(0-∞) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. The placebo group was not evaluated for this outcome measure.
Time Frame: Approximately 96 hours for MK-1006 15mg, 30 mg, 45 mg, 60 mg, 60 mg fed (predose up to approximately 96 hours postdose); approximately 120 hours for MK-1006 80 mg, 100 mg, 140 mg, and 170 mg (predose up to 120 hours postdose)
Population: Participants received a singe dose of MK-1006 following an overnight fast (for approximately 10 hours), except the MK-1006 60 mg fed arm in which participants received a single dose of MK-1006 following the consumption of a standard Japanese breakfast. The same participant may appear in more than one treatment arm.
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5
nM*hr | 489 (134) | 904 (249) | 1900 (384) | 2350 (897) | 2100 (556) | 3820 (1300) | 6060 (2180) | 6920 (1420) | 9560 (3490)
Statistical Analysis 1: Comparison: MK-1006 60 mg vs MK-1006 60 mg Fed; Test type: Superiority or Other; Mixed-effect model; Based on mixed effect model with panel and treatment-within-panel as fixed effects and participant-within panel as a random effect; Geometric mean ratio (fed/fasted) = 0.92

3. Secondary Outcome: Mean Area Under the Plasma Concentration Curve From Time Zero to 24 Hours (AUC[0-24]) After a Single Dose of MK-1006
Description: AUC(0 to 24 hours) was estimated by determining the total area under the curve of the concentration versus time curve to 24 hours post dose. The placebo group was not evaluated for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5
nM*hr | 358 (116) | 665 (186) | 1450 (315) | 1720 (782) | 1440 (342) | 2790 (1000) | 4610 (1730) | 5370 (1330) | 7540 (3010)

4. Secondary Outcome: Mean Maximum Plasma Concentration (Cmax) After a Single Dose of MK-1006
Description: The placebo group was not evaluated for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5
nM | 37.3 (16.3) | 75.4 (23.9) | 169 (49.8) | 185 (102) | 141 (41) | 310 (172) | 514 (180) | 628 (205) | 912 (371)
Statistical Analysis 1: Comparison: MK-1006 60 mg vs MK-1006 60 mg Fed; Test type: Superiority or Other; Mixed-effect model; [statistical method as in outcome 2, analysis 1]; Geometric mean ratio (fed/fasted) = 0.81

5. Secondary Outcome: Median Time to Maximum Plasma Concentration (Tmax) After a Single Dose of MK-1006
Description: The placebo group was not evaluated for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5
hours | 3.0 [2.0 to 5.0] | 4.0 [3.0 to 5.0] | 3.0 [1.0 to 6.0] | 4.0 [1.0 to 5.0] | 5.0 [3.0 to 6.0] | 4.0 [1.0 to 4.0] | 3.5 [1.0 to 6.0] | 5.0 [5.0 to 5.0] | 3.0 [1.0 to 5.0]

6. Secondary Outcome: Apparent Terminal Half-life (T 1/2) After a Single Dose of MK-1006
Description: The apparent half-life was defined as the time required for the plasma concentration of MK-1006 to decrease 50% in the final stage of its elimination. The means and standard deviations displayed as are the harmonic means and pseudo-standard deviations, respectively. The placebo group was not evaluated for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5
hours | 18.0 (5.5) | 18.5 (3.8) | 19.1 (2.2) | 18.5 (3.5) | 17.0 (1.7) | 21.2 (2.9) | 22.1 (5.2) | 20.7 (2.6) | 21.5 (4.0)

7. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: as for outcome 1
Time Frame: up to approximately 17 days
Population: Participants who received study drug. The same participant may appear in more than one treatment arm.
Measure: Number; unit: participants
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg | Placebo | Placebo Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5 | 15 | 2
participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: 24-hour Weighted Mean Glucose (WMG) Concentration
Description: Weighted mean glucose concentration was calculated as the 24-hour area under the plasma concentration-time curve divided by 24.
Time Frame: Up to 36 hours
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg | Placebo | Placebo Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5 | 15 | 2
mg/dL | 206.2 (50.8) [188.0 to 224.4] | 197.6 (40.9) [179.1 to 216.1] | 188.6 (28.0) [170.3 to 206.9] | 178.0 (24.7) [159.5 to 196.6] | 165.7 (26.7) [146.8 to 184.6] | 156.7 (21.7) [138.2 to 175.3] | 199.0 (33.6) [180.7 to 217.3] | 170.4 (25.8) [148.9 to 191.9] | 154.9 (21.4) [134.8 to 175.0] | 214.3 (34.5) [202.9 to 225.7] | 185.4 (17.7) [159.5 to 211.3]
Statistical Analysis 1: Comparison: MK-1006 15 mg vs Placebo; At one or more well tolerated single doses of MK-1006, the 24-hour weighted mean glucose concentration is expected to be at least 25 mg/dL lower than placebo; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; Based on mixed effect model with glucose baseline, panel and treatment-within-panel as fixed effects and participant-within panel as a random effect; Difference in least squares mean = -8.1, 90% CI 2-sided [-23.0 to 6.8] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 15 mg minus LS mean for placebo
Statistical Analysis 2: Comparison: MK-1006 30 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -16.6, 90% CI 2-sided [-32.2 to -1.1] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 30 mg minus LS mean for placebo
Statistical Analysis 3: Comparison: MK-1006 45 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -25.7, 90% CI 2-sided [-40.9 to -10.5] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 45 mg minus LS mean for placebo
Statistical Analysis 4: Comparison: MK-1006 60 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Diffrence in least squares mean = -36.3, 90% CI 2-sided [-52.0 to -20.5] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 60 mg minus LS mean for placebo
Statistical Analysis 5: Comparison: MK-1006 60 mg Fed vs Placebo Fed; Test type: Superiority or Other; p = 0.147, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -19.7, 90% CI 2-sided [-42.2 to 2.7] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 60 mg fed minus LS mean for placebo fed
Statistical Analysis 6: Comparison: MK-1006 60 mg vs MK-1006 60 mg Fed; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = 12.3, 90% CI 2-sided [-0.5 to 25.2] — Difference in least squares mean (LS mean) was calculated as LS mean for MK-1006 60 mg minus LS mean for MK-1006 60 mg fed
Statistical Analysis 7: Comparison: Placebo vs Placebo Fed; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -28.9, 90% CI 2-sided [-49.9 to -7.9] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for placebo fed minus LS mean for placebo
Statistical Analysis 8: Comparison: MK-1006 80 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -57.6, 90% CI 2-sided [-73.3 to -41.9] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 80 mg minus LS mean for placebo
Statistical Analysis 9: Comparison: MK-1006 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -15.3, 90% CI 2-sided [-30.5 to -0.1] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 100 mg minus LS mean for placebo
Statistical Analysis 10: Comparison: MK-1006 140 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -43.9, 90% CI 2-sided [-60.8 to -27.0] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 140 mg minus LS mean for placebo
Statistical Analysis 11: Comparison: MK-1006 170 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — A step down procedure starting with the highest tolerated dose was implemented; [statistical method as in outcome 8, analysis 1]; Difference in least squares mean = -59.4, 90% CI 2-sided [-75.1 to -43.7] — The calculation used to determine the difference in least squares mean (LS mean) was LS mean for MK-1006 170 mg minus LS mean for placebo

ADVERSE EVENTS:
Description: The same participant may appear in more than one treatment arm.
Arm/Group | MK-1006 15 mg | MK-1006 30 mg | MK-1006 45 mg | MK-1006 60 mg | MK-1006 60 mg Fed | MK-1006 80 mg | MK-1006 100 mg | MK-1006 140 mg | MK-1006 170 mg | Placebo | Placebo Fed
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/5 | 0/15 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 0/6 | 1/6 | 1/6 | 3/6 | 1/6 | 1/4 | 1/5 | 1/15 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1006 15 mg (N=6) | MK-1006 30 mg (N=6) | MK-1006 45 mg (N=6) | MK-1006 60 mg (N=6) | MK-1006 60 mg Fed (N=6) | MK-1006 80 mg (N=6) | MK-1006 100 mg (N=6) | MK-1006 140 mg (N=4) | MK-1006 170 mg (N=5) | Placebo (N=15) | Placebo Fed (N=2)
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.